CLINICAL TRIAL: NCT07000331
Title: Effectiveness of Breathing Exercises and Physical Activity Counseling in Individuals Who Have Had COVID-19.
Brief Title: Effectiveness of Exercise and Physical Activity in Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulsah Bargi (Other)
Responsible Party: Sponsor-Investigator, Gulsah Bargi, Principle investigator, Izmir Democracy University
Organization: Izmir Democracy University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Exercise in post-COVID-19
Record Dates: First submitted 2025-05-30; First posted 2025-06-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: physical activity; dyspnea; pain; fatigue; anxiety; depression; quality of life
MeSH Terms: conditions — COVID-19; Motor Activity; Dyspnea; Pain; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind study; the participants were not informed about whether they were in the study group or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The individuals in the study group were given thoracic expansion exercises and physical activity counseling.
  Interventions: Other: Thoracic expansion exercises; Other: Physical activity counseling
- Control group (No Intervention): Individuals in this group continued their normal daily living activities and were followed up only with follow-up.

INTERVENTIONS:
Other: Thoracic expansion exercises — Individuals placed their hands on their lower ribs and then took 3 deep breaths under their hands in a row. After this cycle, individuals rested by taking 3-4 calm breaths. The cycle was repeated 10 times. The individual did this session 4 times a day.
  Arms: Study group
Other: Physical activity counseling — Individuals were given weekly group phone calls and meetings. Individuals were gradually accustomed to regular walking to increase their daily step count. In the first week, individuals were asked to walk a total of 30-45 minutes per day, at least 4-5 days per week, and to increase the number of steps measured at the beginning by approximately 1000-2000 steps per day to reach at least 6500 steps. In the second week, the expected goal was at least 7500 steps. In the third and fourth weeks, they were asked to reach at least 10000 steps.
  Arms: Study group

SUMMARY:
The effects of breathing exercises and physical activity counseling applied for 4 weeks on the number of daily steps, dyspnea, pain, fatigue, mood and quality of life in individuals who have just had COVID-19 are not yet known. For this reason, it was aimed to investigate in this study.

DETAILED DESCRIPTION:
In the COVID-19 pandemic, which deepened the physical inactivity and sedentary lifestyle, the severity and mortality effect of the virus on humans has decreased today. On the other hand, some symptoms may continue to be seen after recovery in individuals who survived COVID-19. It is known that regular physical activities increase immunity and quality of life, reduce stress, anxiety and depression, and support the musculoskeletal and cardiovascular systems. This study aimed to search effects of breathing exercises and physical activity counseling on the step counts, dyspnea, pain, fatigue, mood and quality of life in individuals with post-COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals aged 18 and over who volunteered to participate in the research
* Individuals who can understand and answer surveys
* Compatible individuals who can perform exercises and have good cooperation.
* Individuals who were diagnosed with COVID-19 (individuals with a positive Polymerase Chain Reaction (PCR) test result, compatible with COVID-19 infection as a result of lung X-ray or lung tomography despite negative PCR test results) and discharged after recovery/home quarantine completed

Exclusion Criteria:

* Individuals newly diagnosed with COVID-19, therefore in quarantine at home or receiving treatment in hospital
* Individuals with suspected COVID-19
* Pregnant women
* Individuals with serious psychiatric illness and therefore unable to adapt to exercise sessions
* Individuals with severe cognitive impairment
* Individuals with ongoing orthopedic, neurological, cardiovascular disorders and/or problems which are independent of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Daily step counts | Baseline, at the end of everyday during 4-week and at 4 weeks after baseline evaluation
  Daily average step counts were recorded via a pedometer.

SECONDARY OUTCOMES:
Anxiety score | Baseline and at 4 weeks after baseline evaluation
  The score was obtained from Hospital Anxiety and Depression Scale.The lowest score on this scale is 0 and the highest is 21, with higher scores indicating increased anxiety.
Depression score | Baseline and at 4 weeks after baseline evaluation
  The score was obtained from Hospital Anxiety and Depression Scale.The lowest score on this scale is 0 and the highest is 21, with higher scores indicating increased anxiety.
Dyspnea score | Baseline and at 4 weeks after baseline evaluation
  The score was obtained from Medical Research Council Dyspnea Scale.The lowest score on this scale is 0 and the highest is 4; higher scores indicate increased dyspnea.
Pain score | Baseline and at 4 weeks after baseline evaluation
  The score was obtained from Numerical Rating Scale.The lowest score on this scale is 0 and the highest is 10, with higher scores indicating increased pain.
Fatigue score | Baseline and at 4 weeks after baseline evaluation
  The score was obtained from Numerical Rating Scale.The lowest score on this scale is 0 and the highest is 10, with higher scores indicating increased fatigue.
Quality of life score | Baseline and at 4 weeks after baseline evaluation
  The score was obtained from Short-Form (SF)-36 Quality of life Questionnaire.The lowest score on this scale is 0 and the highest is 100, with higher scores indicating higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Assoc. Dr., Study Director — Izmir Democracy University; SENA UYGUNLAR, Principal Investigator — Izmir Democracy University; GÜLCAN POLAT, Principal Investigator — Izmir Democracy University; DİLAN SU AKTAŞ, Principal Investigator — Izmir Democracy University; UĞUR CANBULAT, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang TJ, Chau B, Lui M, Lam GT, Lin N, Humbert S. Physical Medicine and Rehabilitation and Pulmonary Rehabilitation for COVID-19. Am J Phys Med Rehabil. 2020 Sep;99(9):769-774. doi: 10.1097/PHM.0000000000001505. PMID 32541352
- [Background] Amini H, Isanejad A, Chamani N, Movahedi-Fard F, Salimi F, Moezi M, Habibi S. Physical activity during COVID-19 pandemic in the Iranian population: A brief report. Heliyon. 2020 Nov;6(11):e05411. doi: 10.1016/j.heliyon.2020.e05411. Epub 2020 Nov 2. PMID 33163638